CLINICAL TRIAL: NCT06584825
Title: The Impact of Enhanced Postoperative Vitals Monitoring In-hospital and at Home vs. Standard Care After Inpatient Abdominal and Vascular Surgery: A Pilot Two-centre Randomized Controlled Study
Brief Title: Enhanced Vitals Monitoring After Major Surgery Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Medtronic (Industry); Providence Health Care Ventures (Unknown); Cloud DX Inc. (Industry); Excelar (Unknown); 3D Bridge Solutions (Unknown); Simon Fraser University (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Janny Ke, Anesthesiologist, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H23-03640
Record Dates: First submitted 2024-08-29; First posted 2024-09-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Surgery; Post Operative Complications; Quality of Recovery; General Surgery; Vascular Surgery; Urology; Gynecology
Keywords: Days alive and at home; DAH30; Quality of Recovery 15; Pilot Randomized Controlled Trial; vitals; blood pressure; heart rate; oxygen saturation; device

STUDY DESIGN:
Intervention Model Description: A pilot two-centre randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Vitals Monitoring (Experimental): Enhanced (i.e. additional) monitoring using Health Canada approved devices in-hospital postoperatively, 8am to 5pm from the day of surgery until 3 days after surgery or until discharged (whichever occurs first) followed by twice-daily monitoring at home 3 days after discharge, with a protocol for clinical escalation if vital sign alert thresholds are exceeded.
  Interventions: Device: Enhanced Vitals Monitoring
- Standard Care (No Intervention): Standard vitals monitoring in hospital and standard of care follow-up procedures once discharged home. The research team will administer a questionnaire at 14 and 30 days postoperatively and conduct a 30 day phone call follow-up.

INTERVENTIONS:
Device: Enhanced Vitals Monitoring — For participants in the intervention group, they will receive the enhanced continuous vital sign monitoring, on top of the standard of care monitoring as prescribed per the care team. The enhanced monitoring will be provided during in-hospital postoperatively, 8am to 5pm from the day of surgery until 3 days after surgery or until discharged (whichever occurs first) with a protocol for clinical escalation if vital sign alert thresholds are exceeded, using the Philips monitor (i.e. heart rate and oxygen saturation continuously and blood pressure once an hour while awake). Participants and caregivers will be educated how to put on and off the devices by the study coordinator.
  When participants return home, they will perform twice-daily monitoring using the Cloud DX Inc. Home kit and daily questionnaires at home for 3 days after discharge, with a protocol for clinical escalation if vital sign alert thresholds are exceeded.
  Arms: Enhanced Vitals Monitoring

SUMMARY:
The aim of this clinical trial is to examine the feasibility of an enhanced vital sign monitoring solution in-hospital and at-home. This study includes adult patients undergoing inpatient major vascular or abdominal surgery. Researchers will compare the enhanced vitals monitoring group to the standard of care group to see if it may change post-operative management and outcomes. The primary question it aims to answer is if enhanced monitoring of surgical patient vitals can increase the number of days at home alive in the first 30 days after surgery. Participants in the intervention group will test two vitals monitoring devices, one in the hospital and one at home. They will also be asked to complete several questionnaires and a follow up phone call.

DETAILED DESCRIPTION:
After surgeries, patients are at risk of a variety of complications, thus requiring monitoring for early detection and treatment of complications. The current standard of care consists of continuous monitoring of vital signs during and after anesthetic and/or in the high-acuity and intensive care units, followed by intermittent measurement of vital signs once the patient is in the ward. Once the patient is at home, there is no monitoring nor follow-up.

However, it has been well-established that existing intermittent monitoring of vital signs are too infrequent to capture important vital sign derangements. For example, in an observational study of 312 patients who underwent abdominal surgery, 18% of patients had blood pressure <65 mmHg for at least 15 minutes that were not detected by conventional intermittent monitoring. Nevertheless, it remains unknown the optimal method and duration of increased monitoring for medium-to-high risk surgical patients in-hospital and at home. In a randomized controlled trial (RCT) involving 905 adults undergoing non-elective surgery, remote automated monitoring with virtual care did not reduce the number of days alive and at home 30 days after surgery (DAH30) compared to standard of care. However, there are signals of increased detection of drug errors, decreased pain, and benefits in patients in centres with more escalations in care.

This study is a single-blinded, parallel-group, pilot RCT, with an exploratory feasibility analysis. The study will be reported according to the Consolidated Standards of Reporting Trials (CONSORT) pilot RCT standards.

The study will be conducted at St Paul's Hospital (SPH), Providence Health Care (PHC), in Vancouver, British Columbia, Canada, an academic tertiary care hospital affiliated with the University of British Columbia. The study will also run at and Mount Saint Joseph's (MSJ) Hospital, PHC. The PHC anesthesia and surgical program already has a strong perioperative care focus, featuring enhanced postoperative support available for high risk patients including 1) surgical high-acuity unit (SHAU) with continuous monitoring, run by anesthesiologists, 2) Perioperative Outreach Team that rounds on patients daily for as long as clinically indicated, run by anesthesiologists, 3) multidisciplinary collaboration and support from perioperative internal medicine and/or geriatric teams, with daily rounding for as long as clinically indicated and availability for preoperative consultation and post-discharge follow-up in rapid access clinics, and 4) protocolized monitoring for myocardial injury after non-cardiac surgery for three days according to the Canadian Cardiovascular Society guidelines.

The objective of the study is to obtain pilot data on the enhanced monitoring of vital signs in patients undergoing inpatient major abdominal and/or vascular surgery (i.e. continuous monitoring of vital signs in-hospital (from the day of surgery until 3 days after surgery) followed by twice-daily monitoring at home for 3 days after discharge, with a protocol for care escalation if needed, compared to standard monitoring (intermittent monitoring in-hospital and no monitoring at home).

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing inpatient major abdominal (general surgery, urology, or gynecology) or vascular surgery at St. Paul's Hospital (SPH) and Mount Saint Joseph (MSJ) Hospital
2. Length of stay of at least 48 hours (planned by the clinical team, or by the Canadian Institute of Health Information Discharge Abstract Database Expected Length of Stay (ELOS) for the surgical case mix group
3. Self-reported fluency in reading and speaking in English for patient or home caregiver
4. Living within British Columbia, Canada and in an area that is covered by Bell cellular network (the Cloud DX Inc. device has cellular Long Term Evolution (LTE) using the Bell network).

Exclusion Criteria:

1. Patient refusal
2. Transplant surgery, since these patients have a unique set of considerations and postoperative course.
3. Inability to communicate with research personnel, perform self-monitoring of vital signs, or complete study surveys due to cognitive, language, visual, or hearing barriers
4. Lack of capacity to consent to the study (including under the active influence of sedative medication or having received general anesthetic within the past 24 hours)
5. Unable to use (or does not have a caregiver who can help put on/take off) study monitoring device at home
6. Preoperatively known planned discharge to a nursing home or rehabilitation facility
7. Patient with known allergic reactions to any part material of the device
8. Unable to monitor blood pressure accurately noninvasively using arm blood pressure cuffs, such as due to underlying vascular anatomy or non-pulsatile blood flow physiology
9. Unlikely to be able to return the home monitoring kit (no fixed address, living too far away from site, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Days Alive At Home (DAH30) | Within 30 days after surgery, with the day of surgery as day 0
  Number of days within 30 days of surgery when participants are alive and at home, without visiting an emergency department or urgent care centre or being admitted to a hospital. Home refers to their own home, or a residence of a relative, friend or acquaintance, but excludes a nursing home or a rehabilitation facility.
  If a participant visits an emergency department or urgent care centre, or is admitted to a hospital any time between midnight and 23:59 on a given day, they will lose that day as a day alive at home. If they remain in the care facility past midnight into the next day, then they lose 2 days alive at home. They will continue to lose days alive at home until the day in which they are home from midnight for an entire day. In other words, a day alive at home can be counted only when participants spend an entire day from midnight to 23:59 at home, without being stay at an emergency department, an urgent-care centre or a hospital.

SECONDARY OUTCOMES:
Quality of Recovery at baseline | 14 days after surgery
  Measured using the Quality of Recovery-15 (QoR-15) score. QoR-15 scale is a validated tool to assess the quality of postoperative recovery. It consists of 15 likert questions in two parts.
  Part A consists of 10 questions asking a patient how they have been feeling in the previous 24 hours with regards to factors such as sleeping and eating. Responses are given on an 11 point likert scale from 0 to 10, where 0 is none of the time [poor] and 10 is all of the time [excellent].
  Part B consists of five questions which ask the patient if they have experienced specific adverse events (for example, pain, nausea/vomiting or anxiety). Responses are given on an 11 point likert scale from 10 to 0, where 10 is none of the time [excellent] and 0 is all of the time [poor].
  This questionnaire is administered either over the phone, online or on paper.
Major Morbidity | Within 30 days after surgery, with the day of surgery as day 0
  Complications associated with 30-day mortality: major bleeding, myocardial injury after noncardiac surgery (includes myocardial infarction), myocardial infarction (3rd Universal Definition), sepsis, infection without sepsis, acute kidney injury with new dialysis, stroke, venous thromboembolism and congestive heart failure) within 30 days postoperatively
Mortality | Within 30 days after surgery, with the day of surgery as day 0
  All cause mortality within 30 days of surgery
Emergency Department visit(s) after discharge | Within 30 days after surgery, with the day of surgery as day 0
  This outcome describes if a participant visited an emergency department after discharge within 30 days of surgery, and if so, a count of how many times.
Readmission(s) | Within 30 days after surgery, with the day of surgery as day 0
  This outcome describes if a participant was readmitted to hospital after initial discharge from hospital within 30 days of surgery, and if so, for how long and how many times.
Urgent walk-in clinic visit(s) | Within 30 days after surgery, with the day of surgery as day 0
  This outcome describes if a participant visited an urgent walk-in clinic after discharge within 30 days of surgery, and if so, a count of how many times.
Family doctor clinic visit(s) | Within 30 days after surgery, with the day of surgery as day 0
  This outcome describes if a participant visited a family doctor clinic after discharge within 30 days of surgery, and if so, a count of how many times. This will include details of planned (for suture/staple removal, or other reason) vs. unplanned
Surgeon clinic contact(s) | Within 30 days after surgery, with the day of surgery as day 0
  This outcome describes if a participant visited their surgeon after discharge within 30 days of surgery, and if so, a count of how many times. This will also include details of whether it was a planned (for suture/staple removal, or other reason) vs. unplanned visit and an email, phone call or clinic visit.
Post-Operative Length of Stay | The time from the date of the surgery to the date of discharge from the hospital, up to 30 days after surgery
  The amount of time a patient is in hospital after their operation.
Quality of Recovery at 14 days postoperatively | 14 days after surgery
  Measured using the Quality of Recovery-15 (QoR-15) score. QoR-15 scale is a validated tool to assess the quality of postoperative recovery. It consists of 15 likert questions in two parts.
  Part A consists of 10 questions asking a patient how they have been feeling in the previous 24 hours with regards to factors such as sleeping and eating. Responses are given on an 11 point likert scale from 0 to 10, where 0 is none of the time [poor] and 10 is all of the time [excellent].
  Part B consists of five questions which ask the patient if they have experienced specific adverse events (for example, pain, nausea/vomiting or anxiety). Responses are given on an 11 point likert scale from 10 to 0, where 10 is none of the time [excellent] and 0 is all of the time [poor].
  This questionnaire is administered either over the phone, online or on paper.
Quality of Recovery at 30 days postoperatively | 30 days after surgery with the day of surgery as day 0
  Measured using the Quality of Recovery-15 (QoR-15) score. QoR-15 scale is a validated tool to assess the quality of postoperative recovery. It consists of 15 likert questions in two parts.
  Part A consists of 10 questions asking a patient how they have been feeling in the previous 24 hours with regards to factors such as sleeping and eating. Responses are given on an 11 point likert scale from 0 to 10, where 0 is none of the time [poor] and 10 is all of the time [excellent].
  Part B consists of five questions which ask the patient if they have experienced specific adverse events (for example, pain, nausea/vomiting or anxiety). Responses are given on an 11 point likert scale from 10 to 0, where 10 is none of the time [excellent] and 0 is all of the time [poor].
  This questionnaire is administered either over the phone, online or on paper.

OTHER OUTCOMES:
Completion of the intervention | 30 days after surgery with the day of surgery as day 0
  The primary feasibility outcome is defined as more than 80% of participants completing the monitoring protocol, with a priori definition of the completion being monitoring in-hospital and at home each for 3 times a day for 3 days (or the duration of the hospital stay, whichever is shorter).
Participant Recruitment Rate | Preoperatively, at the time of recruitment, up to 1 month prior to surgery.
  The proportion of patients recruited who provided consent out of all meeting the clinical inclusion criteria
Participant Exclusion Rate | Preoperatively, at the time of screening and recruitment, up to 1 month prior to surgery.
  The proportion of patients excluded out of all patients screened
Participant Withdrawal Rate | Preoperatively, at the time of recruitment, up to 30 days post-operatively
  The proportion of patients who withdrew from the study out of all enrolled patients.
Participant patterns of use of monitoring devices | Up to 30 days after surgery, with the day of surgery as day 0
  How frequently did patients use the monitoring devices and for what duration. This will be based on data collected from the devices. The monitoring will take place for 3 days after surgery in hospital, or until discharge (whichever occurs first) and 3 days once the patient returns home.
Device issues encountered | Up to 30 days after surgery, with the day of surgery as day 0
  Issues that participants reported encountering with the monitoring devices. Reported as an open ended question in the patient daily log sheet
Reasons for device removal | Up to 30 days after surgery, with the day of surgery as day 0
  What were the reasons that patients took the monitors on and off (e.g. charging/battery life, showers, eating, mobilization/physiotherapy) as reported as an open ended question in the patient daily log sheet
Interruptions in vitals monitoring | Up to 30 days after surgery, with the day of surgery as day 0
  Description of instances of interruption in monitoring that were more than 4 hours
In-Hospital Enhanced Monitoring Device System Usability Scale | At the time of discharge from hospital or 3 days after surgery (whichever occurs first)
  Patient feedback about enhanced monitoring device usability of the in-hospital enhanced monitoring device. The System Usability Scale (SUS) is a patient-reported measurement which includes ten 5-point likert scale questions from 1 to 5, with one being strongly disagree and 5 being strongly agree. The suitability of using SUS for evaluating medical devices has been well established.
At-Home Enhanced Monitoring Device System Usability Scale | Between 3 days after hospital discharge to 30 days after surgery, with the day of surgery as day 0
  Patient feedback about enhanced monitoring device usability of the at-home enhanced monitoring devices. The System Usability Scale (SUS) is a patient-reported measurement which includes ten 5-point likert scale questions from 1 to 5, with one being strongly disagree and 5 being strongly agree. The suitability of using SUS for evaluating medical devices has been well established.
Care escalation frequency | Up to 30 days after surgery, with the day of surgery as day 0
  The frequency of vital sign derangements detected by enhanced monitoring and the resulting care escalation categorized by type of vital measure within the duration of monitoring. This will be determined based on data from the devices and as reported by the patients nurse.
Response time | Up to 30 days after surgery, with the day of surgery as day 0
  Time between vital sign alert and care escalation. This will be determined based on data from the devices and as reported by the patients nurse.
  xii. logistics of device use (time spent on education, initiation, discontinuation, cleaning, collection, and troubleshooting of devices) xiii. issues that arise in the workflow
Logistics of Enhanced Monitoring Implementation | Up to 30 days after surgery, with the day of surgery as day 0
  Description of the logistics of implementing the intervention. This includes a description of time spent on education, initiation, discontinuation, cleaning, collection, and troubleshooting of the devices by the study coordinator.
Workflow Issues | Up to 30 days after surgery, with the day of surgery as day 0
  A qualitative description of issues that arise in the workflow of implementing the intervention.
Adverse Events | Up to 30 days after surgery, with the day of surgery as day 0
  Any patient-reported adverse events
Patient Feedback | 30 days after surgery, with the day of surgery as day 0
  An evaluation of potential harm or safety issues gathered from a feedback questionnaire filled out by the participant at the end of the enhanced monitoring period. The Feedback questionnaire uses a 5 point likert scale (1-5), where 1 = Strongly disagree…3 = Neutral…5 = Strongly agree. The questionnaire asks patients to rate how they feel about the following statements:
  i. Their ability to move around after surgery ii. Their daily activities (e.g. going to the bathroom, eating, showering) iii. Making them anxious about your health? There is also one open ended question for participants to add any other feedback they have related to enhanced monitoring
Study Costs | Pre-study and up to time of publication
  Overall study costs spent and difference of costs between intervention group and standard care group
Questionnaire Completion | From time of enrollment to 30 days after surgery with the day of surgery as day 0
  Completion rates of all questionnaires administered
Method of Questionnaire Completion | From time of enrollment to 30 days after surgery with the day of surgery as day 0
  Number of participants that completed questionnaires over the phone, online or on paper.
Support needed for questionnaires | From time of enrollment to 30 days after surgery with the day of surgery as day 0
  Number of participants that required either caregiver or family member or technical support to complete questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Janny Ke, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Mount Saint Joseph's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT06584825/Prot_SAP_000.pdf